CLINICAL TRIAL: NCT04083313
Title: Analysis of Endoloops, Endostaples and Endoclips for Closing the Appendiceal Stump During Laparoscopic Appendectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Mislav Rakić, MD, Head of the Department of Hepatobilliary surgery, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UHDubrava1
Record Dates: First submitted 2019-08-26; First posted 2019-09-10 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Appendicitis Acute; Laparoscopic Surgery
Keywords: Laparoscopic appendectomy; Endoloop; Endostapler; Endoclip
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Endoloop (Active Comparator): Patients in which appendiceal stump was ligated using Endoloop
  Interventions: Device: Technique used for closing the appendiceal stump
- Endostapler (Active Comparator): Patients in which appendiceal stump was ligated using Endostapler
  Interventions: Device: Technique used for closing the appendiceal stump
- Endoclip (Active Comparator): Patients in which appendiceal stump was ligated using Endoclip
  Interventions: Device: Technique used for closing the appendiceal stump

INTERVENTIONS:
Device: Technique used for closing the appendiceal stump — In all patients, laparoscopic appendectomy is performed, only difference is the way of managing appendiceal stump
  Other Names: Laparoscopic appendectomy

SUMMARY:
In this randomized control trial the patients with acute appendicitis will be divided in three groups according to the management of the appendiceal stump(Endostapler, Endoloop or Endoclip). Pre-, peri- and postoperative data will be analysed.

DETAILED DESCRIPTION:
Acute appendicitis is the most common indication for intraabdominal emergency surgery, and appendectomy is one of the most commonly performed procedures in abdominal surgery. Today laparoscopic appendectomy (LA) has the status of a ''Gold Standard'' treatment, and it is accepted as the treatment of choice for acute appendicitis.There are several ways of closing the appendiceal stump.An inadequate closure of the appendiceal stump can lead to morbidity of operated patients. The aim of this study is to assess the efficiency of different closure techniques by focusing on the intraoperative and postoperative complications.The patients will be divided into three groups based on the technique used for appendiceal stump closure, whether it is Endoloop, Endostapler or Endoclip. In the patients included in the study the investigators will analyse demographic data, peroperative laboratory values, clinical data and treatment outcomes. Also, the histopathological findings of the specimens and perioperative and postoperative complications will be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically and radiologically(Ultrasound) verified appendicitis

Exclusion Criteria:

* Patients converted from laparoscopy to open surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Operative and postoperative complications | Seven postoperative days
  Number of all complications will be presented in total numbers.
Operative and postoperative complications | Seven postoperative days
  Complications will be presented as a percentage of the all operated patients.

SECONDARY OUTCOMES:
Value levels of leukocytes | Before surgery
  Whit blood cells count
Duration of symptoms | Before surgery
  Duration of symptoms will be measured in hours.
Height | Before surgery
  Meters
Weight | Before surgery
  Kilograms
C-reactive protein | Before surgery
  Milligrams/liter
Neutrophiles | Before surgery
  Neutrophile count
Body mass index | Before surgery
  Kilograms/meter square
Body temperature | Before surgery
  Body temperature will be measured in degrees celsius.
Length of the operations | During operation
  Length of the operations will be presented in minutes.
Closure of the appendiceal stump using Endoloop | During operation
  Number of patients in which this technique was performed.
Closure of the appendiceal stump using Endoloop | During operation
  Percentage of the all operated patients in which this technique was used.
Closure of the appendiceal stump using Endostapler | During operation
  Number of patients in which this technique was performed
Closure of the appendiceal stump using Endostapler | During operation
  Percentage of the all operated patients in which this technique was used.
Closure of the appendiceal stump using Endoclip | During operation
  Number of patients in which this technique was performed
Closure of the appendiceal stump using Endoclip | During operation
  Percentage of the all operated patients in which this technique was used.
Number of reoperated patients | Seven days
  Presented in total numbers
Hospital stay | Seven days
  Length of the hospital stay will be presented in days.
Histopathological findings | Seven days
  Histopathological findings will be graduated in 3 grades - phlegmonous,gangrenous and perforated.
Percentage of reoperated patients | Seven days
  Presented in percentages

CONTACTS AND LOCATIONS:
Locations (1):
- UH Dubrava, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaghoubian A, Kaji AH, Lee SL. Laparoscopic versus open appendectomy: outcomes analysis. Am Surg. 2012 Oct;78(10):1083-6. PMID 23025946
- [Background] Rashid A, Nazir S, Kakroo SM, Chalkoo MA, Razvi SA, Wani AA. Laparoscopic interval appendectomy versus open interval appendectomy: a prospective randomized controlled trial. Surg Laparosc Endosc Percutan Tech. 2013 Feb;23(1):93-6. doi: 10.1097/SLE.0b013e318277df6a. PMID 23386160
- [Background] Beldi G, Muggli K, Helbling C, Schlumpf R. Laparoscopic appendectomy using endoloops: a prospective, randomized clinical trial. Surg Endosc. 2004 May;18(5):749-50. doi: 10.1007/s00464-003-9156-z. Epub 2004 Mar 19. PMID 15026904
- [Background] Beldi G, Vorburger SA, Bruegger LE, Kocher T, Inderbitzin D, Candinas D. Analysis of stapling versus endoloops in appendiceal stump closure. Br J Surg. 2006 Nov;93(11):1390-3. doi: 10.1002/bjs.5474. PMID 16862615
- [Background] Wagner M, Aronsky D, Tschudi J, Metzger A, Klaiber C. Laparoscopic stapler appendectomy. A prospective study of 267 consecutive cases. Surg Endosc. 1996 Sep;10(9):895-9. doi: 10.1007/s004649900192. PMID 8703146
- [Background] Safavi A, Langer M, Skarsgard ED. Endoloop versus endostapler closure of the appendiceal stump in pediatric laparoscopic appendectomy. Can J Surg. 2012 Feb;55(1):37-40. doi: 10.1503/cjs.023810. PMID 22269300